CLINICAL TRIAL: NCT00459979
Title: A Phase II Study of Sunitinib Malate in Patients With Renal Cell Carcinoma and Unresectable Primary Tumors
Brief Title: Sunitinib in Treating Patients With Kidney Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE17806; P30CA043703 (NIH); CASE-17806 (Other: Case Comprehensive Cancer Center); CASE-17806-CC209 (Other: Cancer Center IRB)
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; stage III renal cell cancer; stage IV renal cell cancer; papillary renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental)
  Interventions: Drug: sunitinib malate; Procedure: conventional surgery

INTERVENTIONS:
Drug: sunitinib malate — Sunitinib will be dosed at 50 mg p.o. daily
  Other Names: SUNITINIB L-Malate salt; SU010398; PHA-290940AD; Sutent; SUNITINIB
Procedure: conventional surgery — nephrectomy

SUMMARY:
RATIONALE: Sunitinib may stop the growth of kidney cancer by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying the side effects and how well sunitinib works in treating patients with kidney cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the percentage of patients with renal cell carcinoma and unresectable primary tumors who can achieve sufficient tumor response, according to the operating surgeon, to undergo nephrectomy after sunitinib therapy.
* To evaluate the safety of sunitinib in patients with renal cell carcinoma and unresectable primary tumors, including analysis of the morbidity of surgery after sunitinib therapy
* To evaluate the objective response rate of patients with renal cell carcinoma and unresectable primary tumors who receive sunitinib therapy.

OUTLINE: A single arm phase II study of sunitinib in patients with unresectable renal cell carcinoma (RCC) will be conducted, including patients with and without distant metastases.

Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 42 days in the absence of disease progression or unacceptable toxicity. Surgery is performed if and when primary tumor becomes resectable. Patients with residual and/or metastatic disease may resume sunitinib malate within 8 weeks after surgery.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 31 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal cell carcinoma (any histology) based on prior biopsy or biopsy performed and reviewed at Cleveland Clinic Foundation. This can include pathology read as adenocarcinoma consistent with renal origin.
* Unresectable primary tumor due to any of the following factors or various combinations thereof:

  * Large tumor size (> 15 cm)
  * Bulky lymphadenopathy (> 4 cm or encasement of renal vessels or great vessels)
  * Venous thrombosis (high level/invasive disease requiring inferior vena cava reconstruction or hypothermic circulatory arrest)
  * Proximity to vital structures (e.g., mesenteric vasculature)
  * Any one of these factors may or may not constitute unresectability, but for consideration for this trial, the surgical and medical oncologist must agree that the particular constellation of findings for the patient under consideration would likely entail a low probability (<50%) that the tumor would be resectable (with negative margins) or that the potential morbidity associated with an attempt at surgical resection would not be clinically acceptable. The numerical thresholds noted above are only a guideline and the clinical judgment of the surgeon and medical oncologist will determine unresectability.
* Patients with history of brain metastases can be enrolled 2 weeks following the completion of gamma knife or whole brain radiotherapy.
* ECOG performance status (PS) 0-1 or Karnofsky PS >/=70%
* Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 times upper limit of normal (ULN)
* Total Serum Bilirubin ≤ 1.5 times ULN
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)
* Serum calcium ≤ 12.0 mg/dL
* Creatinine ≤ 2.5 mg/dL
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* The presence of any of the following will exclude a patient from study enrollment:
* Prior systemic treatment for RCC.
* Evidence of bleeding diathesis or coagulopathy. Patients with hematuria from the primary renal tumor are eligible provided all other eligibility criteria are met.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, severe peripheral vascular disease (claudication) or procedure on peripheral vasculature, coronary/peripheral artery bypass graft, New York Heart Association grade II or greater congestive heart failure, cerebrovascular accident or transient ischemic attack, clinically significant bleeding or pulmonary embolism.
* Hypertension that cannot be controlled by medications to < 160/90 mmHg.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Pregnancy or breastfeeding.
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2011-03 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian I. Rini, MD, Study Chair — Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Lane BR, Derweesh IH, Kim HL, O'Malley R, Klink J, Ercole CE, Palazzi KL, Thomas AA, Rini BI, Campbell SC. Presurgical sunitinib reduces tumor size and may facilitate partial nephrectomy in patients with renal cell carcinoma. Urol Oncol. 2015 Mar;33(3):112.e15-21. doi: 10.1016/j.urolonc.2014.11.009. Epub 2014 Dec 19. PMID 25532471
- [Derived] Rini BI, Garcia J, Elson P, Wood L, Shah S, Stephenson A, Salem M, Gong M, Fergany A, Rabets J, Kaouk J, Krishnamurthi V, Klein E, Dreicer R, Campbell S. The effect of sunitinib on primary renal cell carcinoma and facilitation of subsequent surgery. J Urol. 2012 May;187(5):1548-54. doi: 10.1016/j.juro.2011.12.075. Epub 2012 Mar 14. PMID 22425095

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: sunitinib malate : Sunitinib will be dosed at 50 mg p.o. daily
  conventional surgery : nephrectomy
Period: Overall Study
Arm/Group | Sunitinib
Started | 30
Completed | 28
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: Years]
  Median age | 61 (10.0) [37 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Response to Sunitinib Therapy
Description: Defined as a reduction in tumor burden to such an extent that nephrectomy is permitted within 1 year of the start of therapy. No response to sunitinib therapy is defined as a nephrectomy not being permitted within 1 year of the start of therapy or removal from the study for any reason
Time Frame: 1 year from start of treatment
Population: per protocol - analysis after at least one cycle of Sunitinib
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 28
participants | 13

2. Secondary Outcome: The Number of Patients With Any Type of Complication or Adverse Event
Description: The safety of sunitinib will be assessed by recording the number of patients with any type of complication or adverse event within 1 year of the start of therapy.
Time Frame: 1 year from start of treatment
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 28
participants | 28

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the amount of time (in months) between the start of treatment and documented RECIST defined progression. RECIST progression is defined as at least a 20% increase in the sum of diameters of target lesions, in addition to an absolute increase of at least 5mm.
Time Frame: 1 year from start of treatment
Measure: Median (Full Range); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 28
months | 11.2 [1.7 to 36.5]

4. Secondary Outcome: Percent Decrease of Diameter of Primary Tumors
Description: Median percent decrease in size in all primary renal cell carcinoma tumors. Response was unconfirmed by RECIST criteria because patients went to surgery and did not undergo follow-up scans.
Time Frame: 1 year from start of treatment
Population: per protocol - analysis after at least one cycle of Sunitinib
Measure: Median (Full Range); unit: percentage of tumors diameter decrease
Units Other Than Participants: tumors
Arm/Group | Sunitinib
Number analyzed (Participants) | 28
Number analyzed (tumors) | 35
percentage of tumors diameter decrease | 22 [-13 to 100]

5. Secondary Outcome: Number of Tumors Which Decreased in Size
Description: Number of tumors with at least some reduction in longest primary tumor diameter. Response was unconfirmed by RECIST criteria because patients went to surgery and did not undergo follow-up scans.
Time Frame: 1 year from start of treatment
Population: per protocol - after at lease one cycle of Sunitinib
Measure: Number; unit: tumors
Units Other Than Participants: tumors
Arm/Group | Sunitinib
Number analyzed (Participants) | 28
Number analyzed (tumors) | 35
tumors | 28

6. Secondary Outcome: Number of Tumors With 30% Reduction in Size
Description: Number of tumors with at least 30% reduction in longest primary tumor diameter. Response was unconfirmed by RECIST criteria because patients went to surgery and did not undergo follow-up scans.
Time Frame: 1 year from start of treatment
Population: per protocol- after at least one cycle of Sunitinib
Measure: Number; unit: tumors
Units Other Than Participants: tumors
Arm/Group | Sunitinib
Number analyzed (Participants) | 28
Number analyzed (tumors) | 35
tumors | 13

7. Secondary Outcome: Median Size Reduction Among Tumors With Some Shrinkage
Description: The median size reduction in the largest diameter of the primary RCC tumor among the tumors with at least some shrinkage in diameter
Time Frame: 1 year from start of treatment
Measure: Median (Full Range); unit: cm
Units Other Than Participants: tumors with size reduction
Arm/Group | Sunitinib
Number analyzed (Participants) | 28
Number analyzed (tumors with size reduction) | 28
cm | 1.6 [0.4 to 5.1]

ADVERSE EVENTS:
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 16/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=28)
Hemoglobin (Blood and lymphatic system disorders) | 4
Platelets (Blood and lymphatic system disorders) | 1
Supraventricular and nodal arrhythmia - Atrial fibrillation (Blood and lymphatic system disorders) | 2
Cardiac ischemia/infarction (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Perforated Bowel (Gastrointestinal disorders) | 1
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 1
Hemorrhage, GU - Urinary NOS (Reproductive system and breast disorders) | 3
Hemorrhage, pulmonary/upper respiratory - Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 3
"Pain - NOS (General disorders) | 1
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2
Obstruction, GU - Bladder (Renal and urinary disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=28)
Hemoglobin (Blood and lymphatic system disorders) | 17
Leukocytes (total WBC) (Investigations) | 12
Lymphopenia (Investigations) | 4
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 12
Platelets (Investigations) | 22
Hypertension (Vascular disorders) | 14
Hypotension (Vascular disorders) | 4
Constitutional Symptoms - Other (Specify, __) (General disorders) | 5
Fatigue (asthenia, lethargy, malaise) (General disorders) | 24
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2
Insomnia (General disorders) | 3
Weight loss (General disorders) | 4
Cheilitis (Skin and subcutaneous tissue disorders) | 4
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 9
Hypopigmentation (Skin and subcutaneous tissue disorders) | 6
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 8
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 19
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 13
Anorexia (Gastrointestinal disorders) | 16
Constipation (Gastrointestinal disorders) | 18
Dehydration (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 23
Distension/bloating, abdominal (Gastrointestinal disorders) | 2
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 3
Heartburn/dyspepsia (Gastrointestinal disorders) | 12
Hemorrhoids (Gastrointestinal disorders) | 6
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 7
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 17
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 12
Hematoma (Vascular disorders) | 2
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 2
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 6
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 5
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 8
Hemorrhage, pulmonary/upper respiratory - Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 3
Hemorrhage/Bleeding - Other (Vascular disorders) | 2
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 3
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 7
Infection with unknown ANC - Dental-tooth (Infections and infestations) | 2
Infection with unknown ANC - Pharynx (Infections and infestations) | 4
Edema: head and neck (Blood and lymphatic system disorders) | 4
Edema: limb (Blood and lymphatic system disorders) | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3
Alkaline phosphatase (Investigations) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 9
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 12
Bilirubin (hyperbilirubinemia) (Investigations) | 3
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2
Creatinine (Investigations) | 11
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6
Uric acid, serum-high (hyperuricemia) (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 10
Neuropathy: sensory (Nervous system disorders) | 3
Syncope (fainting) (Nervous system disorders) | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 9
Pain - Back (Musculoskeletal and connective tissue disorders) | 4
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 2
Pain - Dental/teeth/peridontal (Gastrointestinal disorders) | 2
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 12
Pain - Head/headache (Nervous system disorders) | 8
Pain - Joint (Musculoskeletal and connective tissue disorders) | 5
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 4
Pain - Oral cavity (Gastrointestinal disorders) | 3
Pain - Other (Specify, __) (General disorders) | 2
Pain - Rectum (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 3
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes